## Development of methods and algorithms for diet design based on gut microbiota analysis

## Statistical analysis

Number of clinical trial: 1631

**Project number: NSP67** 

Approved by Ethical Committe of National Institute for Health Development 25.10.2016

## Statistical analysis

Based on sample size calculations, we estimated that with 17 participants, the study would have more than 80% power to detect a significant difference among weight loss study group, assuming a mean BMI reduction by 3 kg/m2, with a mean BMI and standard deviation of 35 and 3.2 kg/m2, respectively, at an alpha level of 5%.

Statistical analysis included bacteria with average colonization frequency > 70% and average abundance > 0.001. Analysis of data was carried out in R statistical programming language, version 3.5.0 (28). The resulting p-values were corrected for multiple comparisons for each phylogenetic level using Benjamini-Hochberg correction (FDR). A corrected p-value < 0.1 was considered statistically significant. Unless stated otherwise, corrected P values are shown in the text.

Pairwise comparisons were evaluated using Wilcoxon signed-rank test, for the comparison of test and reference groups Kruskal-Wallis test was applied.

To control for within-subject variability, we used the subsequent sample-pairs as within-subject controls and compared  $\beta$ -diversity before and after the intervention. This was also applied to reference group samples. The following cutoffs were used: \*, p < 0.05; \*\*, p < 0.01; \*\*\*\*, p < 0.001; \*\*\*\*\*, p < 0.0001.

## Agglomerative hierarchical clustering

Ward's agglomerative hierarchical clustering on a distance matrix was generated from a species by sample Bray-Curtis distance matrix. The method produces a dendrogram by treating each sample as a singleton cluster, merging pairs of clusters until all clusters have been merged into one big cluster containing all samples. Ward's agglomeration method minimizes the total within-cluster variance.